CLINICAL TRIAL: NCT02548455
Title: A Clinical Evaluation of the Safety of the St. Jude Medical Quartet 1457Q Left Ventricular Lead, an IDE Study
Brief Title: Quartet 1457Q Left Ventricular (LV) Lead Investigational Device Exemption (IDE) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRD 616
Record Dates: First submitted 2015-09-10; First posted 2015-09-14 (Estimated); Results first posted 2018-05-08 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment (Experimental): Subjects implanted with the Quartet 1457Q LV lead
  Interventions: Device: Quartet 1457Q LV Lead

INTERVENTIONS:
Device: Quartet 1457Q LV Lead

SUMMARY:
The primary intent of this study is to assess the safety of the model 1457Q Quartet LV lead at 3 months in a patient population indicated for cardiac resynchronization therapy.

DETAILED DESCRIPTION:
This is a prospective, multi-center, IDE clinical study designed to evaluate the safety of the Model 1457Q Quartet LV lead.

A minimum of 94 and a maximum of 430 subjects will be enrolled in this study at up to 40 centers worldwide.

All subjects successfully implanted with a Quartet 1457Q lead will be followed every 6 months post implant until Pre Market Approval (PMA) is obtained or the study is closed.

ELIGIBILITY:
Inclusion Criteria:

1. Meets current St. Jude Medical clinical indication for implantation of a cardiac resynchronization therapy system:

   " to provide a reduction of the symptoms of moderate to severe heart failure (New York Heart Association Functional Class III or IV) in those patients who remain symptomatic despite stable, optimal medical therapy and have a left ventricular ejection fraction ≤ 35% and a prolonged QRS duration, OR " to maintain synchrony of the left and right ventricles in patients who have undergone an Atrio Ventricular nodal ablation for chronic (permanent) atrial fibrillation and have New York Heart Association Functional Class II or III heart failure.
2. Is receiving a new market-approved St. Jude Medical quadripolar cardiac resynchronization therapy system implant with the Quartet 1457Q LV lead.
3. Have the ability to provide informed consent for study participation and is willing and able to comply with the prescribed follow-up tests and schedule of evaluations.
4. Are 18 years or above, or of legal age to give informed consent specific to state and national law.

Exclusion Criteria:

1. Had a previous unsuccessful commercial or non-Quartet 1457Q LV lead implant attempt
2. Have a hypersensitivity to a single 1.0mg dose of dexamethasone sodium phosphate
3. Patient is currently participating or plans to participate in a potentially confounding drug or device trial during the course of this study. Co-enrollment in other studies may be allowed if pre-approval is granted from the study manager.
4. Are pregnant or planning pregnancy in the next 6 months
5. Have a life expectancy of less than 24 months due to any condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 499 (Actual)
Dates: Start 2015-10-27 (Actual); Primary Completion 2016-08-19 (Actual); Study Completion 2017-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Delurgio, MD, Study Chair — Emory University
Locations (30):
- United States (30):
  - Heart Center Research, Huntsville, Alabama
  - Arizona Arrhythmia Research Center, Phoenix, Arizona
  - Cardiology Associates of Northeast Arkansas, Jonesboro, Arkansas
  - Scripps Health, La Jolla, California
  - Premier Cardiology, Inc., Newport Beach, California
  - Stanford University Hospital, Stanford, California
  - Munroe Regional Medical Center, Ocala, Florida
  - Tallahassee Research Institute, Tallahassee, Florida
  - Emory University Hospital, Atlanta, Georgia
  - North Georgia Heart Foundation, Gainesville, Georgia
  - Iowa Heart Center, West Des Moines, Iowa
  - Central Baptist Hospital, Lexington, Kentucky
  - One Health Cardiology, Owensboro, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Thoracic Cardiovascular Healthcare Foundation, Lansing, Michigan
  - Missouri Heart Center, Columbia, Missouri
  - Catholic Medical Center, Manchester, New Hampshire
  - Cardiovascular Associates of Delaware Valley, Haddon Heights, New Jersey
  - Forsyth Medical Center, Winston-Salem, North Carolina
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Oklahoma Heart Institute at Utica, Tulsa, Oklahoma
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Donald Guthrie Foundation for Education & Research, Sayre, Pennsylvania
  - Greenville Health System, Greenville, South Carolina
  - Erlanger Medical Center, Chattanooga, Tennessee
  - The Stern Cardiovascular Foundation, Germantown, Tennessee
  - The Heart Hospital Baylor Plano, Plano, Texas
  - Swedish Medical Center - Heart & Vascular, Seattle, Washington
  - St. Mary's Hospital, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: Left Ventricular Lead model Quartet 1457Q
  Left Ventricular Lead
Period: Overall Study
Arm/Group | Treatment
Started (484 were successful and 15 were unsuccessful.) | 499 (A total of 499 subjects were enrolled at 31 investigational sites.)
Completed Pre-Discharge | 484
Completed 6-Month Follow-up | 259
Completed 12-Month Follow-up | 61 (Study completed prior to all subjects reaching the 6- and 12-month visits.)
Completed | 259 (Completed 6-Month Follow-up)
Not Completed | 240
Not completed — Withdrawal by Subject | 27
Not completed — Death | 26
Not completed — Lost to Follow-up | 14
Not completed — Visit not completed | 173

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 499
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.3 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 194
  Male | 305
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 491
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 39
  White | 450
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 499

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Free From LV Lead-related Complications Through 3 Months
Description: A complication is defined as a Serious Adverse Device Effect related to the Quartet 1457Q lead. A Serious Adverse Device Effect is an event related to the use of a medical device that led to death, a life-threatening illness or injury, a permanent impairment to a body structure or a body function, an in-patient or prolonged hospitalization, medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to a body structure or a body, a malignant tumor OR fetal distress, fetal death or a congenital abnormality or birth defect.
Time Frame: 3 months
Population: The first 94 subjects who underwent an attempted implant of the Quartet 1457Q lead and either completed a 3-month follow-up visit, withdrew from the study or died prior to the 3-month follow-up visit.
Measure: Count of Participants; unit: Participants
Groups:
- Treatment: Subjects implanted with the Quartet 1457Q left ventricular lead
Arm/Group | Treatment
Number analyzed (Participants) | 94
Participants | 4
Statistical Analysis 1: Comparison: Treatment; The hypothesis for the endpoint is: H0: Freedom from LV lead-related complications through 3 months (91 days) ≤ 85% H1: Freedom from LV lead-related complications through 3 months (91 days) > 85% A total of 85 subjects were required to have at least 80% power to reject the null hypothesis at the 5% significance level at three months (91 days) post-implant or attempted implant. After accounting for 9% attrition, the required sample size was 94 subjects; Test type: Equivalence — Freedom from left ventricular lead-related complications through 3 months was estimated to be 96.0% with a 95% lower confidence bound of 92.6% based on the Promote Q IDE study (NCT00990665), and 98.3% with a 95% lower confidence bound of 97.7% based on data from the Quadripolar Post-Approval study (NCT01555619); p = 0.05, Log Rank; Kaplan-Meier Estimate = 85

ADVERSE EVENTS:
Time Frame: Adverse event data was collected on all subjects from enrollment through 12 months of follow-up.
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 27/499
Serious Adverse Events (participants affected / at risk) | 60/499
Other Adverse Events (participants affected / at risk) | 56/499
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=499)
Cardiac Tamponade (Injury, poisoning and procedural complications) | 3 (3)
Coronary Sinus Dissection (Injury, poisoning and procedural complications) | 4 (4)
Coronary Sinus Perforation (Injury, poisoning and procedural complications) | 1 (1)
Excessive Bleeding (Injury, poisoning and procedural complications) | 2 (2)
Hematoma/Seroma (Injury, poisoning and procedural complications) | 1 (1)
Induced Arrhythmias Atrial/Ventricular (Injury, poisoning and procedural complications) | 2 (2)
Infections (Injury, poisoning and procedural complications) | 1 (1)
Infections (Infections and infestations) | 5 (5)
Lead Dislodgement (Injury, poisoning and procedural complications) | 20 (20)
Lead Dislodgement (Product Issues) | 14 (14)
Loss of Pacing/Sensing (Product Issues) | 1 (1)
Pectoral/Diaphragmatic Stimulation (Injury, poisoning and procedural complications) | 1 (1)
Pericardial Effusion (Injury, poisoning and procedural complications) | 1 (1)
Pneumothorax (Injury, poisoning and procedural complications) | 6 (6)
Pulmonary Edema (Injury, poisoning and procedural complications) | 2 (2)
Rise in Threshold (Injury, poisoning and procedural complications) | 1 (1)
Rise in Threshold (Product Issues) | 1 (1)
Anesthesia Complication (Injury, poisoning and procedural complications) | 1 (1)
Cardiogenic Shock (Injury, poisoning and procedural complications) | 1 (1)
Elevated Pacing Threshold (Injury, poisoning and procedural complications) | 1 (1)
Guide Wire Problem (Injury, poisoning and procedural complications) | 1 (1)
Hypotension (Injury, poisoning and procedural complications) | 1 (1)
Loose Set Screw (Injury, poisoning and procedural complications) | 1 (1)
Respiratory Compromise (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper Extremity Deep Vein Thrombosis (Injury, poisoning and procedural complications) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=499)
Cardiac/Coronary Sinus Dissection (Injury, poisoning and procedural complications) | 2 (2)
Cardiac/Coronary Sinus Perforation (Injury, poisoning and procedural complications) | 1 (1)
Hematoma/Seroma (Injury, poisoning and procedural complications) | 7 (7)
Induced Atrial or Ventricular Arrythmias (Injury, poisoning and procedural complications) | 1 (1)
Infection (Injury, poisoning and procedural complications) | 1 (1)
Lead Dislodgement (Injury, poisoning and procedural complications) | 5 (6)
Lead Dislodgement (Product Issues) | 1 (1)
Local Tissue Reaction; Formation of Fibrotic Tissue (Skin and subcutaneous tissue disorders) | 1 (1)
Pectoral/Diaphramatic/Phrenic Nerve Stimulation (Injury, poisoning and procedural complications) | 20 (22)
Pectoral/Diaphramatic/Phrenic Nerve Stimulation (Product Issues) | 10 (10)
Oversensing (General disorders) | 2 (2)
Upper Extremity Discomfort (Injury, poisoning and procedural complications) | 1 (1)
Oversensing (Injury, poisoning and procedural complications) | 1 (1)
Should Pain (Injury, poisoning and procedural complications) | 1 (1)
Suture Sleeve Disruption (Injury, poisoning and procedural complications) | 1 (1)
Upper Extremity Deep Vein Thrombosis (Injury, poisoning and procedural complications) | 3 (3)
Device Reset Mode (Product Issues) | 1 (1)
Elevated Threshold (Product Issues) | 1 (1)
Oversensing (Product Issues) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less